CLINICAL TRIAL: NCT00004365
Title: Study of Pituitary Size and Function in Familial Dwarfism of Sindh
Status: Completed | Type: Observational
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: Northwestern University (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Other Study IDs: 199/11940; NU-571
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-12

CONDITIONS: Growth Hormone Deficiency
Keywords: endocrine disorders; growth hormone deficiency; rare disease
MeSH Terms: conditions — Dwarfism, Pituitary; Endocrine System Diseases; Rare Diseases

SUMMARY:
OBJECTIVES: I. Assess pituitary size and anatomic configuration by magnetic resonance imaging (MRI) in 4 affected dwarfs in the province of Sindh, Pakistan.

II. Evaluate ultradian growth hormone (GH) secretory patterns in 4 affected dwarfs.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: Pituitary size and anatomy and growth hormone response are evaluated.

All patients undergo MRI of the pituitary fossa on day 1. On day 2, homozygous patients receive a slow infusion of normal saline with blood sampling every 10 minutes.

ELIGIBILITY:
* Familial Dwarfism of Sindh
* Severe short stature but proportionate without dysmorphic features
* Normal body size and weight at birth
* Bone age is severely delayed
* Puberty is somewhat delayed (age 15-16)
* Fertility present in at least 3 dwarfs

Ages: 10 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4
Dates: Start 1995-09; Study Completion 2000-02

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Baumann, Study Chair — Northwestern University

REFERENCES:
- [Background] Baumann G, Maheshwari H. The Dwarfs of Sindh: severe growth hormone (GH) deficiency caused by a mutation in the GH-releasing hormone receptor gene. Acta Paediatr Suppl. 1997 Nov;423:33-8. doi: 10.1111/j.1651-2227.1997.tb18366.x. PMID 9401536
- [Background] Maheshwari HG, Silverman BL, Dupuis J, Baumann G. Phenotype and genetic analysis of a syndrome caused by an inactivating mutation in the growth hormone-releasing hormone receptor: Dwarfism of Sindh. J Clin Endocrinol Metab. 1998 Nov;83(11):4065-74. doi: 10.1210/jcem.83.11.5226. PMID 9814493